CLINICAL TRIAL: NCT03340350
Title: Minocycline for Treatment of Posttraumatic Stress Disorder in Veterans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sriram Ramaswamy (U.S. Federal Agency)
Collaborators: Creighton University (Other)
Responsible Party: Sponsor-Investigator, Sriram Ramaswamy, Staff Psychiatrist, VA Nebraska Western Iowa Health Care System
Organization: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAM-01068
Record Dates: First submitted 2017-06-06; First posted 2017-11-13 (Actual); Results first posted 2020-06-17 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: PTSD
Keywords: Minocycline; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minocycline (Experimental): Minocycline 100 mg/day 1 to 7 and 200 mg/day 8 to end of week 12
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline capsule
  Other Names: Minocycline hydrochloride capsule

SUMMARY:
The study will evaluate the safety and efficacy of adjunctive minocycline treatment in veterans with PTSD.

DETAILED DESCRIPTION:
This is a 12-week, open-label pilot study in which adjunctive minocycline will be administered to approximately 15 veterans diagnosed with PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans between the ages of 19 and 65 who meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for chronic PTSD.
2. Patients who have been taking an adequate dose of selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) medication, bupropion, or mirtazapine for a minimum of 8 weeks at the time of study entry.
3. PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) score of > 33 at the Screening Visit. Eligible persons will be allowed to have other symptoms that are commonly comorbid with PTSD (e.g., anxiety, somatic symptoms). This strategy will provide a feasible and generalizable sample of those with chronic PTSD.

Exclusion Criteria:

1. Patients with a concurrent DSM-5 diagnosis in any of the following categories:

   1.1. Major Neurocognitive Disorder (NCD) 1.2. Lifetime Schizophrenia and other Psychotic Disorders 1.3. Lifetime Bipolar Disorder 1.4. Alcohol Dependence or Abuse in 3 months prior to the Screening Visit 1.5. Any other Substance Dependence or Abuse (excluding nicotine) in 12 months prior to the Screening Visit 1.6. Any other concurrent Axis I Disorder (including Major Depressive Disorder) must be secondary to the primary diagnosis of PTSD.
2. Chronic pain levels requiring use of any opiate medications with the exception of Tramadol. Patients are allowed the use of Tramadol at 25-50 mg per day dosing.
3. Any condition or disorder that may cause neuropsychiatric sequelae (e.g., Parkinson's disease, stroke, seizures, or TBI).
4. Past chronic PTSD, meaning PTSD that preceded the incident traumatic event responsible for the current PTSD. Other traumatic life events will not be exclusionary unless they resulted in previous PTSD.
5. Patients with a history of intolerance or hypersensitivity to minocycline or other tetracycline antibiotics, or prior tetracycline use 2 months prior to the Screening Visit.
6. Concomitant treatment with penicillin or other antibiotics, or treatment with antibiotics for greater than 7 days in the past month.
7. Use of aspirin, non-steroidal anti-inflammatory agents (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors for < 6 months prior to study entry or dose changes after study entry. Limited as-needed use is permitted prior to study entry but not during the study.
8. Use of statins will not be permitted during the study as they have been shown to reduce levels of pro-inflammatory cytokines.
9. Use of concomitant anti-coagulant drugs (except low-dose aspirin) as minocycline has been shown to depress plasma prothrombin activity.
10. Any degree of hepatic or renal failure that in the Investigator's judgement would pose a safety risk for treatment with minocycline.
11. Conditions which may be negatively affected by minocycline treatment, such as active inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease).
12. A history of C. difficile colitis.
13. Patients who based on history or mental status examination have a significant risk of committing suicide, or who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
14. Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
15. Women who are pregnant or plan to become pregnant during the study. All women of childbearing potential must have a negative urine pregnancy test at the Screening Visit and throughout the study. Sexually active women participating in the study must use a medically acceptable form of contraception.
16. Patients with a current known infection or who are acutely ill.
17. Patients with an autoimmune disease (i.e., Lupus, Rheumatoid Arthritis).
18. Immunocompromised patients (i.e., HIV).
19. Patients with thyroid disorders unless euthyroid at screening.
20. Patients with cancer not in remission.
21. Patients with cardiovascular disease, such as myocardial infarction and arrhythmias.
22. Patients with diabetes.
23. History of significant esophagitis.
24. Patients who plan to initiate or terminate any psychotropic medication during the study. Patients taking any psychotropic medication should be on a stable dose for at least 6 weeks prior to the Screening Visit (except for the SSRI, SNRI or mirtazapine used to treat their PTSD) AND agree not to discontinue or otherwise alter treatment during the study.
25. Patients who plan to initiate or terminate any form of psychotherapy or behavior therapy during the study with the exception of PTSD Orientation Group. Subjects may be in supportive psychotherapy if it was initiated at least three months prior to the Screening Visit AND subject agrees not to discontinue or otherwise alter therapy during the study. Subjects receiving evidence-based psychotherapies such as Prolonged Exposure or Cognitive Processing Therapy will be excluded.
26. Patients who are unable to speak, read, and understand English or are judged by the Investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, MD, Principal Investigator — VA Nebraska Western Iowa Health Care System
Locations (1):
- VA Nebraska-Western Iowa Health Care System, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline
Started | 10
Completed | 4
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6
  Black | 1
  Hispanic or Latino | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptom Severity
Description: PTSD symptom severity was assessed using total scores on the Past Month version of the Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (CAPS-5). Total scores on the CAPS-5 range from 0 to 80, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Minocycline: Participants received minocycline 100 mg/day 1 to 7 and 200 mg/day 8 to end of week 12
  Minocycline: Minocycline capsule
Arm/Group | Minocycline
Number analyzed (Participants) | 4
score on a scale
  Baseline | 31.5 (7.23)
  Week 12 | 23 (7.62)

2. Primary Outcome: Change in C-reactive Protein (CRP) Level
Description: Measure of inflammation
Time Frame: Screening and Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Minocycline
Number analyzed (Participants) | 4
mg/dL
  Screening | 1.25 (0.35)
  Week 12 | 0.90 (0.14)

3. Primary Outcome: Change in Interleukin 6 (IL-6) Level
Description: Measure of inflammation
Time Frame: Screening and Week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Minocycline
Number analyzed (Participants) | 4
pg/mL
  Screening | 1.27 (0.49)
  Week 12 | 1.64 (0.67)

4. Primary Outcome: Change in Tumor Necrosis Factor Alpha (TNF-α) Level
Description: Measure of inflammation
Time Frame: Screening and Week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Minocycline
Number analyzed (Participants) | 4
pg/mL
  Screening | 1.14 (0.31)
  Week 12 | 1.13 (0.14)

5. Secondary Outcome: Depression Symptom Severity
Description: Depression symptom severity was assessed using total scores on the Beck Depression Inventory-II (BDI-II). Total scores on the BDI-II range from 0 to 63, with higher scores indicating greater severity of depression symptoms.
Time Frame: Screening and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline
Number analyzed (Participants) | 4
score on a scale
  Screening | 24.5 (12.71)
  Week 12 | 20.75 (5.19)

6. Secondary Outcome: Clinical Status (Severity)
Description: The Clinical Global Impressions Severity scale (CGI-S) was used to assess severity of illness. Scores on the CGI-S range from 0 to 7, with higher scores reflecting greater severity of illness.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline
Number analyzed (Participants) | 4
score on a scale
  Baseline | 4.25 (0.50)
  Week 12 | 4.00 (0.00)

7. Secondary Outcome: Clinical Status (Improvement)
Description: The Clinical Global Impressions Improvement scale (CGI-I) was used to assess global improvement in clinical status. Scores on the CGI-I range from 0 to 7, with lower scores reflecting greater improvement in clinical status.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline
Number analyzed (Participants) | 4
score on a scale
  Baseline | 4.00 (0.00)
  Week 12 | 3.25 (0.96)

8. Secondary Outcome: Executive Functioning (Set Shifting)
Description: The Trail Making Test (TMT) is a scale used to measure a type of executive functioning (i.e., higher-order cognitive function) called set shifting. The TMT is scored as time (in seconds) to complete Parts A and B of this task. A difference score was calculated (time to complete Part B minus time to complete Part A) to subtract the motor component of this task and provide a better estimate of executive functioning. Lower difference scores on the TMT indicate better set shifting.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Minocycline
Number analyzed (Participants) | 4
seconds
  Baseline | 43.75 (11.62)
  Week 12 | 23.00 (1.92)

9. Secondary Outcome: Executive Functioning (Verbal Fluency)
Description: The Controlled Oral Word Association (COWA) is a scale used to measure a type of executive functioning (i.e., higher-order cognitive function) called verbal fluency. The COWA is scored as the total number of valid words produced in one minute for each of three letters, with 1 point scored for each valid word (score range: 0-no upper limit). Higher scores on the COWA indicate greater verbal fluency.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Minocycline
Number analyzed (Participants) | 4
number of words
  Baseline | 31.00 (4.00)
  Week 12 | 32.25 (6.65)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Minocycline
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=10)
Rash/hives (Skin and subcutaneous tissue disorders) | 2
Hospitalization (General disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT03340350/Prot_SAP_000.pdf